CLINICAL TRIAL: NCT02635438
Title: "A Multi-Centre, Randomized, Double Blind, Parallel-Group, Comparative Clinical Trial to Evaluate the Safety and Clinical Equivalence of Generic Clotrimazole Troche/Lozenges USP, 10mg (Unique Pharmaceutical Laboratories, India) to Clotrimazole Troche/Lozenges ® 10mg (Roxane Laboratories Inc., USA) in Subjects With Oropharyngeal Candidiasis ".
Brief Title: A Comparative Clinical Trial to Evaluate the Safety and Clinical Equivalence of Clotrimazole Troche/Lozenges USP, 10mg (Unique Pharmaceutical Laboratories, India) With Clotrimazole Troche 10mg (Roxane Laboratories Inc., USA) in Subjects With Oropharyngeal Candidiasis.
Acronym: TPC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thinq Pharma-CRO Pte. Ltd. (Industry)
Collaborators: Unique Pharmaceuticals Ltd, India (Unknown); THINQ Pharma CRO Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPC-CLT-002
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Oropharyngeal Candidiasis
Keywords: Oropharyngeal Candidiasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Test Product: Clotrimazole troche/ lozenges USP, 10 mg (Unique Pharmaceutical Laboratories, India) 10mg troche 5 times a day for 14 consecutive days
  Interventions: Drug: Unique Pharmaceutical Laboratories, India
- Arm B (Active Comparator): Reference Product: Clotrimazole Troche/Lozenges ® 10mg (Roxane Laboratories Inc., USA) troche 5 times a day for 14 consecutive days
  Interventions: Drug: Roxane Laboratories Inc., USA

INTERVENTIONS:
Drug: Unique Pharmaceutical Laboratories, India — Clotrimazole troche/ lozenges, 10 mg 5 times a day for 14 consecutive days
  Arms: Arm A
Drug: Roxane Laboratories Inc., USA — Clotrimazole Troche/ Lozenges USP, 10 mg 5 times a day for 14 consecutive days
  Arms: Arm B

SUMMARY:
The objectives of this study are to compare the efficacy and safety of Clotrimazole troche/ lozenges USP, 10 mg (Unique Pharmaceutical Laboratories, India) vs. Clotrimazole Troche/ Lozenges USP, 10 mg (Roxane Laboratories Inc., USA) in patients with oropharyngeal candidiasis, where this condition has been diagnosed by clinical examination and confirmed by fungal culture

DETAILED DESCRIPTION:
This study is Randomized, Double Blind, Parallel, Comparative study. Approximately 26 study sites across India will participate in this study to complete sample size of 360 randomized subjects in order to achieve at least 250 per-protocol (PP) subjects.

Subjects would be assigned randomly to test product or reference product in 1:1 ratio.

Subjects with confirmed oral candidiasis by KOH smear/candidal culture will be given study medication 5 times a day for 14 consecutive days.

The schedule of the subject's visit at study site will be as follows:

1. Visit 1 - Screening visit (-7 Days).
2. Visit 2 - Randomization (Day 1).
3. Visit 3 - Follow Up (Day 8 (+2)).
4. Visit 4 - Follow Up (Day 15 (+2)).
5. Visit 5 - Follow Up/ End of study (Day 21 (+/-4)) Subjects with complete resolution of signs and symptoms of Oral Candidiasis on Day 21 (+/-4) will be considered as treatment success.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of specific signs and symptoms of Oropharyngeal Candidiasis, including erythematous areas, white patches(thrush), mouth pain, irritation, burning, glossitis, altered taste, pruritis, dysphagia and odynophagia.
2. Clinical examination of oropharynx consistent with a diagnosis of oral candidiasis (such as creamy, white, curd-like patches of "thrush" or erythematous lesions on mucosal surfaces).
3. Confirmation of Candidiasis by findings on direct microscopic examination (potassium hydroxide smear) consistent with Candida species or positive fungal culture for Candida species, with culture obtained in the 2 days preceding initiation of therapy with the study drug.
4. Subjects who are able and willing to give Informed Consent.

Exclusion Criteria:

1. Female subjects who are pregnant, lactating or planning to become pregnant during the study period.
2. Subjects diagnosed with disseminated candidiasis or requiring systemic antifungal therapy.
3. Subjects diagnosed with hairy leukoplakia.
4. Presence of only perioral lesions, e.g., angular chelitis.
5. History of intolerance or sensitivity to clotrimazole (or other imidazole or azole compounds) or any constituent of Roxane ® or the generic Clotrimazole Troche/ Lozenges or unable to tolerate oral medication.
6. Subjects having history of resistance to treatment with clotrimazole (Subject who are resistant to Clotrimazole after culture and sensitivity test have to be excluded from the study).
7. Subjects who have received any oral or systemic antifungal therapy within fourteen (14) days prior to randomization.
8. Subjects who have received any investigational therapy within 30 days prior to randomization.
9. Subjects who have been diagnosed with any concomitant condition that, in the opinion of the investigator, could interfere with the evaluation of efficacy or safety, or would make it unlikely that the subject would complete the study.
10. Subjects who have been treated with protease inhibitors for the first time within 30 days.
11. Subjects who have been taking medications known to have significant interaction with azoles (e.g., antacids, H2-receptor blockers, rifampin, phenytoin, carbamazepine, astemizole).
12. Subjects who have a history of candidal prophylaxis with any azole antifungal medication.
13. Any subject with recurrent Oropharyngeal Candidiasis.
14. Any subject who is chronically infected with Candida.
15. Any subject with baseline liver function tests greater than 3 times the upper limit of normal (ULN).
16. CD4 cell count less than 200 cells/mm3. 17. Absolute neutrophil count less than 500/mm3.

18. Subject with history of Type II Diabetes Mellitus with Uncontrolled Blood Sugar levels. (I.e. Random Blood Sugar level > 350).

19. Suspected inability (or) unwillingness to comply with the study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Clinical Cure | 7 days after the end of the therapy, (Day 21(+/- 4)
  Clinical cure i.e., complete resolution of all signs and symptoms of Oropharyngeal Candidiasis, 7 days after the end of the therapy, (Day 21(+/- 4)). Signs and Symptoms of Oral Candidiasis will be assessed using the Murray scale on day 21(+/- 4). According to the Murray Scale, lesion score 0 and symptom score 0 is considered as clinical cure.

SECONDARY OUTCOMES:
Mycological Cure | Day 15(+2) of therapy.
  Mycological cure (negative culture and negative KOH for Candida species) at Day 15(+2) of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Kumar, Medical, Study Director — Director Medical Services, Unique Pharmacutical Laboratories, India (A Division Of J. B. Chemicals and Pharmacuticals Limited)
Locations (26):
- India (26):
  - Grant Government Medical College & Sir JJ group of Hospital, Mumbai, Maharashtra
  - Curie Manavata Cancer Centre, Nashik, Maharashtra
  - Manas Hospital, Nashik, Maharashtra
  - Gujrat Cancer and Research Institute, Ahmadābād
  - HCG Hospital, Ahmadābād
  - Sujan Surgical Cancer Hospital & Amravati cancer foundation, Amravati
  - Dr Hedgewar Hospital, Aurangabad
  - Maulana Azad Medical College, Delhi
  - Bhagwan Mahaveer Cancer Hospital and Research Centre, Jaipur
  - Chittaranjan National Cancer Institute, Kolkata
  - Saroj Gupta Cancer Centre & Research Institute, Kolkata
  - Mandya institute of medical science, Mandya
  - Father Muller Medical College Hospital, Mangalore
  - Tata Memorial Hospital, Mumbai
  - Government Medical Colllege Nagpur, Nagpur
  - Shree hospital and critical care centre, Nagpur
  - Sir Ganga Ram Hospital, New Delhi
  - Ashwin Medical Foundations Moraya Multispeciality Hospital, Pune
  - Deenanath Mangeshkar Hospital and Research Centre, Pune
  - P.D.E.AS Ayurved Rugnalaya & Sterling Multispeciality Hospital, Pune
  - Rajiv Gandhi Institute of Medical Science and RIMS Government Hospital, Srikakulam
  - Apple Hospital, Surat
  - Asian Institute of Medical Science, Thane
  - Kailash cancer hospital and research center, Vadodara
  - Medical College and S.S.G Hospital, Vadodara
  - S.B.K.S. Medical Institute & Research Centre, Vadodara